CLINICAL TRIAL: NCT04120753
Title: A Multi-center, Randomized, Open-label, Active-controlled, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of OLOMAX Tab in Hypertension Patients With Low-Intermediate Risk for Cardiovascular Disease
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of OLOMAX Tab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1351_P401
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — olmesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment 1 (Experimental): OLOMAX 20/5/5mg
  Interventions: Drug: OLOMAX 20/5/5mg
- Treatment 2 (Experimental): OLOMAX 20/5/10mg
  Interventions: Drug: OLOMAX 20/5/10mg
- Treatment 3 (Active Comparator): Olmesartan 20 mg/Amlodipine 5 mg
  Interventions: Drug: Olmesartan 20 mg/Amlodipine 5 mg

INTERVENTIONS:
Drug: OLOMAX 20/5/5mg — Tablets, Oral, QD
  Other Names: Olomax Tablet
  Arms: Treatment 1
Drug: OLOMAX 20/5/10mg — Tablets, Oral, QD
  Other Names: Olomax Tablet
  Arms: Treatment 2
Drug: Olmesartan 20 mg/Amlodipine 5 mg — Tablets, Oral, QD
  Other Names: Sevikar HCT
  Arms: Treatment 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of OLOMAX Tab (20/5/5mg, 20/5/10mg) in Hypertension Patients with Low-Intermediate Risk for Cardiovascular Disease.

DETAILED DESCRIPTION:
The patients who meet the inclusion/exclusion criteria will be randomized 1:1:1 to test group 1 (olomax tablet 20/5/5mg), test group 2 (olomax tablet 20/5/10mg), and control group (sevica tablet 5/20mg.

After randomization, the drug will be administered for 8 weeks according to the assigned group.

During the administration period, subjects will conduct a total of three outpatient visits at 4 weeks (Visit 3) and 8 weeks (Visit 4, EOS), including randomized visits (Visit 2).

ELIGIBILITY:
Inclusion Criteria:

Screening (Visit 1) Inclusion Criteria

1. Men and women over 19 years of age as of the date of written consent
2. High blood pressure patients who meet the following criteria - In case of new arrivals, Sitting systolic blood pressure (sitSBP) ≥ 160 mmHg or sitting diastolic blood pressure (sitDBP) ≥ 100 mmHg, or

   * If you are taking one antihypertensive drug from the Angiotensin II Receptor Blocker (ARB) or Calcium-Channel Blocker (CCB) class, sitSBP ≥ 140 mmHg or sitDBP ≥ 90 mmHg, or
   * If you are taking ARB and CCB class antihypertensive drugs together
3. Those who meet the following mLDL-C criteria* (*Korean Society of Lipid and Atherosclerosis Dyslipidemia Treatment Guideline 3)

   - For cardiovascular disease low risk group #1, LDL-C ≥ 130 mg/dL or
   * For intermediate risk group #2 for cardiovascular disease, LDL-C ≥ 100 mg/dL. #1: Low-risk group: Those who do not have the following major cardiovascular risk factors other than high blood pressure

     #2: Moderate risk group: People with one or more of the following major cardiovascular risk factors other than hypertension
   * Age (men ≥45 years, women ≥55 years)
   * Family history of early onset coronary artery disease (coronary artery disease occurs in family members [parents, siblings] <55 years old for men and <65 years old for women)
   * Smoking
   * High density lipoprotein-cholesterol (HDL-C) <40 mg/dL (However, in case of HDL-C ≥60 mg/dL, 1 is subtracted from the number of major risk factors.)
4. Those who voluntarily agree to participate in clinical trials and sign a written consent form

Random allocation (visit 2) Inclusion criteria

1. Those who have medication compliance of more than 70% during the introduction period of Sevica Tablet 5/20 mg and have good TLC performance according to the investigator's judgment
2. Those who meet the following test values for each institution at the time of the baseline (visit 2) visit ① For low-risk cardiovascular disease group, mLDL-C ≥ 130 mg/dL or For those at moderate risk for cardiovascular disease, mLDL-C ≥ 100 mg/dL

Exclusion Criteria:

* Patient with hypersensitivity Olmesartan, Amlodipine, Rosuvastatin, dihydropyridine
* Who disagreed to perform effective contraception during the clinical trial
* Orthostatic hypotension with symptoms
* Secondary hypertension and suspected secondary hypertension
* Creatinine clearance < 30mL/min
* AST(Aspartate Aminotransferase) or ALT(Alanine Aminotransferase) level ≥ 3x ULN (upper limit of normal range)

  1. Patients with hypersensitivity to the main ingredient (Olmesartan, Amlodipine or Rosuvastatin) or components of the investigational drug or dihydropyridine derivatives
  2. Pregnant and lactating women, women and men of childbearing potential who do not agree to use appropriate contraception during the clinical trial period

     * Implantation of an intrauterine device or intrauterine system, ② Double barrier method for men or women of childbearing potential (condoms and contraceptive diaphragms, vaginal sponges or cervical caps), ③ Sterilization procedures (vasectomy, bilateral tubal ligation, etc.)
  3. Patients with symptomatic orthostatic hypotension
  4. Patients with secondary hypertension or patients suspected of having secondary hypertension (e.g. aortic coarctation, hyperaldosteronism, renal artery stenosis, Cushing's syndrome, pheochromocytoma, polycystic kidney disease, etc.)
  5. Those with confirmed medical history, concomitant diseases, or surgical history/procedure history:

     ① The following cardiovascular disease occurred within 24 weeks from the time of screening
* Coronary artery disease, atherosclerotic ischemic stroke and transient cerebral ischemic attack, peripheral artery disease, carotid artery disease (limited to cases where significant carotid artery stenosis is confirmed), abdominal aneurysm, severe aortic stenosis, coronary artery revascularization (PTCA or CABG) , Arrhythmias requiring treatment (ventricular tachycardia, etc.)

  * Myopathy, including rhabdomyolysis, that occurred within 24 weeks from the time of screening

    ③ Biliary obstruction occurring within 24 weeks from the time of screening
    * Severe liver failure that occurred within 24 weeks from the time of screening ⑤ Drug or alcohol abuse within 1 year from the time of screening ⑥ Major mental illness (depression, bipolar disorder, etc.) ⑦ Malignant tumor within 5 years from the time of screening 6) Persons confirmed to have abnormalities in the following laboratory tests at the time of screening and randomization ① CK ≥ 2
  * Triglyceride (TG) ≥ 500 mg/dL ③ Active liver disease including persistent ALT elevation of unknown cause or AST ≥ 3 ④ The following renal function abnormalities:
* Kidney dialysis or
* Patients with severe renal impairment (creatinine clearance (CLcr) < 30 mL/min)

  * Hyperkalemia (K >5.5 mEq/L)

    * Hyponatremia (Na <135 mEq/L) or uncorrected sodium depletion ⑦ Hyperuricemia (Uric acid >10 mg/dL) 7) Those who have taken statin drugs or non-statin lipid regulators within 8 weeks before screening 8) Those expected to be administered the following drugs during the clinical trial period, including screening

      * Aliskiren ② Cyclosporine ③ Statin preparations other than clinical investigational drugs ④ Vistatin lipid regulators other than clinical investigational drugs
  * Antihypertensive drugs other than clinical investigational drugs ⑥ Other drugs that may affect blood lipids 9) People with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption 10) A person who has received another investigational drug or a clinical trial medical device within 30 days before screening 11) Other people deemed unsuitable for participation in clinical trials according to the judgment of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
mLDL-C change rate (%) | 8 weeks
  mLDL-C change rate (%) at 8 weeks after administration compared to baseline in test group 1 and control group
mLDL-C change rate | 8 weeks
  mLDL-C change rate (%) at 8 weeks after administration compared to baseline in test group 2 and control group

SECONDARY OUTCOMES:
Change rate (%) in mLDL-C | 4 weeks
  Change rate (%) in mLDL-C at 4 weeks of administration of investigational drug compared to baseline
cLDL-C* change rate | 4 weeks
  cLDL-C* change rate (%) at 4 weeks of administration of investigational drug compared to baseline
cLDL-C* change rate | 8 weeks
  cLDL-C* change rate (%) at 8 weeks of administration of investigational drug compared to baseline
Change amount and rate of change (%) in each of the following lipid indicators | 4 weeks
  Change amount and rate of change (%) in each of the following lipid indicators at 4 weeks of administration of the investigational drug compared to the baseline
Change amount and rate of change (%) in each of the following lipid indicators | 8 weeks
  Change amount and rate of change (%) in each of the following lipid indicators at 8 weeks of administration of the investigational drug compared to the baseline
Proportion of test subjects with mLDL-C less than 70 mg/dL | 4 weeks
  Proportion of test subjects with mLDL-C less than 70 mg/dL at 4 weeks of administration of investigational drug (%)
Proportion of test subjects with mLDL-C less than 70 mg/dL | 8 weeks
  Proportion of test subjects with mLDL-C less than 70 mg/dL at 8 weeks of administration of investigational drug (%)
Proportion of test subjects with mLDL-C less than 100 mg/dL | 4 weeks
  Proportion of test subjects with mLDL-C less than 100 mg/dL at 4 weeks of administration of investigational drug (%)
Proportion of test subjects with mLDL-C less than 100 mg/dL | 8 weeks
  Proportion of test subjects with mLDL-C less than 100 mg/dL at 8 weeks of administration of investigational drug (%)
Change and rate of change in sitSBP (%) | 4 weeks
  Change and rate of change in sitSBP (%) at 4 weeks of administration of investigational drug compared to baseline
Change and rate of change in sitDBP (%) | 8 weeks
  Change and rate of change in sitDBP (%) at 8 weeks of administration of investigational drug compared to baseline
Blood pressure normalization* rate (% | 8 weeks
  Blood pressure normalization* rate (%) at 8 weeks after administration of investigational drug
Change amount and rate of change (%) | 4 weeks
  Change amount and rate of change (%) in each of the following sugar indicators at 4 weeks of administration of the investigational drug compared to the baseline
Change amount and rate of change (%) | 8 weeks
  Change amount and rate of change (%) in each of the following sugar indicators at 8 weeks of administration of the investigational drug compared to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Inho Chae, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Daewoong pharmatceutical, Seoul, South Korea

REFERENCES:
- [Derived] Kim BJ, Cha KS, Cho WH, Kim EJ, Choi SH, Kim MH, Kim SH, Park JB, Park SM, Sohn IS, Ryu KH, Chae IH. Efficacy and Safety of a Single-Pill Triple Combination of Olmesartan, Amlodipine, and Rosuvastatin in Hypertensive Patients with Low-to-Moderate Cardiovascular Risk: A Multicenter, Randomized, Open-Label, Active-Control, Phase IV Clinical Trial. J Cardiovasc Pharmacol Ther. 2023 Jan-Dec;28:10742484231205204. doi: 10.1177/10742484231205204. PMID 37814541